CLINICAL TRIAL: NCT01543594
Title: Study of Efficacy and Safety of Biologic Drugs in the Therapy of Rheumatoid Arthritis and Spondyloarthritis
Brief Title: Italian Registry of Arthritis on Biologic Therapy
Acronym: GISEA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Studio Early Arthritis (Network)
Responsible Party: Principal Investigator, Prof. Florenzo Iannone, Associate Professor of Rheumatology, University of Bari, Gruppo Italiano Studio Early Arthritis
Other Study IDs: DG-624; 2012 (Other: ANMAR)
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Seronegative polyarthritis; Biologic drugs; Safety efficacy biologics polyarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The biologic drugs targeting TNFa, IL-6, IL-1, T cells, B cells have represented a fundamental discovery to treat rheumatic patients whose disease appears to be refractory to conventional therapy. These biologic drugs have been registered for human therapy from a few years, thereby the investigators miss long-term data for safety and efficacy. Aim of this study is to register all the clinical data of patients with rheumatoid arthritis and spondyloarthritis beginning a treatment with biologic drugs in order to assess the long-term safety and efficacy in the real life.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Rheumatoid arthritis, Ankylosing spondylitis, Psoriatic arthritis
* Patients with active disease refractory to traditional disease modifying drugs (methotrexate, leflunomide, sulphasalazine, cyclosporine, hydrossiclorochine)
* Patients eligible to begin conventional biologic therapy

Exclusion Criteria:

* Any criteria excluding treatment with biologic drugs according to international guidelines

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by active polyarthritis beginning conventional biologic drugs
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2009-01; Primary Completion 2022-05 (Estimated); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Florenzo Iannone, MD, Study Chair — University of Bari
Locations (1):
- GISEA, Bari, Italy

REFERENCES:
- [Derived] Cacciapaglia F, Manfredi A, Erre G, Piga M, Sakellariou G, Viapiana O, Gremese E, Spinelli FR, Atzeni F, Bartoloni E. Correspondence on 'Characteristics associated with hospitalisation for COVID-19 in people with rheumatic disease: data from the COVID-19 global rheumatology alliance physician-reported registry' by Gianfrancesco M et al. The impact of cardiovascular comorbidity on COVID-19 infection in a large cohort of rheumatoid arthritis patients. Ann Rheum Dis. 2023 Jul;82(7):e159. doi: 10.1136/annrheumdis-2020-218813. Epub 2020 Sep 15. No abstract available. PMID 32933920
- [Derived] Iannone F, La Montagna G, Bagnato G, Gremese E, Giardina A, Lapadula G. Safety of etanercept and methotrexate in patients with rheumatoid arthritis and hepatitis C virus infection: a multicenter randomized clinical trial. J Rheumatol. 2014 Feb;41(2):286-92. doi: 10.3899/jrheum.130658. Epub 2014 Jan 15. PMID 24429167